CLINICAL TRIAL: NCT03274206
Title: A Phase 2b Trial to Evaluate the Efficacy and Safety of BLS-ILB-E710c in Patients With Cervical Intraepithelial Neoplasia 2/3 (CIN2/3)
Brief Title: A Trial to Evaluate the Efficacy and Safety of BLS-ILB-E710c in Patients With Cervical Intraepithelial Neoplasia 2/3 (CIN2/3)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioLeaders Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLS-ILB-E710c-202; 12591 (Other: Ministry of Food and Drug Safety)
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3
Keywords: Cervical Intraepithelian Neoplasia Grade 2/3; CIN 2/3; HPV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BLS-ILB-E710c (Experimental): * Drug: BLS-ILB-E710c 1,000mg
  * Dosage and duration: 4 capsules per day for 5 consecutive days at week 1,2,4, and 8)
  Interventions: Biological: BLS-ILB-E710c
- BLS-ILB-E710c-placebo (Placebo Comparator): * Drug: BLS-ILB-E710c-placebo
  * Dosage and duration: 4 capsules per day for 5 consecutive days at week 1,2,4, and 8)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: BLS-ILB-E710c — BLS-ILB-E710c 250mg/capsule
  Arms: BLS-ILB-E710c
Drug: Placebo — BLS-ILB-E710c-placebo
  Arms: BLS-ILB-E710c-placebo

SUMMARY:
This study evaluates the efficacy and safety of the experimental drug, BLS-ILB-E710c, in patients with Cervical Intraepithelial Neoplasia 2/3 (CIN2/3). 2/3 of participants will receive the experimental drug, while 1/3 of participants will receive placebo.

DETAILED DESCRIPTION:
Primary Outcome Measure:

Complete histopathological regression from baseline [Time Frame: Baseline through Week 16]

Secondary Outcome Measures:

* Change from baseline of CIN classification [Time Frame: Baseline through Week 16]
* Change from baseline of RCI [Time Frame: Baseline through Week 16 and Week 32]
* Change from baseline of cytopathological classification based on bethesda system [Time Frame: Baseline through Week 16 and Week 32]
* Change from baseline as compared to placebo in the expression rate of P16/Ki-67 [Time Frame: Baseline through Week 16]
* Change from baseline as compared to placebo of the number of CD8 positive cells in the cervical tissue [Time Frame: Baseline through Week 16]
* Change from baseline as compared to placebo in HPV 16 clearance rate
* Change of RCI based on the histopathological regression at Week 16 [Time Frame: Week 16 through Week 32]

ELIGIBILITY:
Inclusion Criteria:

* Fertile female aged between 20 and 49
* Subjects who are infected with HPV 16 type only or with HPV 16 type and any other types listed below

  1) low risk type of HPV, 2) HPV 16-related type
* Subjects who are diagnosed as Cervical interaepithelial neoplasia 2/3 (CIN2/3) by colposcopic biopsy within 6 weeks before enrollment
* All lesions must be observable by colposcopy and CIN2 or higher lesion must be less than 1/2 in the transformation zone area
* Willing to use adequate contraception methods during the study period
* Eligible based on screening test results
* Normal electrocardiogram
* Voluntarily signed informed consent form

Exclusion Criteria:

* Subjects who are diagnosed with Carcinoma In Situ with microinvasion or suspicious invation
* Presence of adenocarcinoma or glandular lesion in the cervix
* Subjects who are infected with HPV type 18-related type
* Subjects with autoimmune disease
* Current or prior treatment past 2 months with immunosuppressant therapies
* Hypersensitive to the investigational drug
* Subjects who currently have acute diseases that require medical attention
* Participation in other studies involving investigational drug(s) or investigational device(s) within 3 months
* Currently having chronic pancreatitis or diagnosed with acute pancreatitis
* Currently having underlying diseases including inflammatory intestinal diseases and tumors, ulcer, bleeding or puncture in the gastrointestinal tract
* Pregnant or breastfeeding
* Subjects with active or inactive hepatitis, or infectious disease
* History of HIV infection
* History of therapeutic HPV vaccination
* Subjects who require continuous use of antibiotics
* Administration of blood product within 3 months before signing informed consent form
* History of vaccination within 2 months before signing informed consent form (4 months in case of live vaccine)

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Regression rate | Baseline through Week 16
  The rate of complete histopathological regression from baseline as compared to placebo

SECONDARY OUTCOMES:
CIN classification | Baseline through Week 16
  Change from baseline of CIN classification
Change of Reid's Colposcopic Index (RCI) | Baseline through Week 16 and Week 32
  Change from baseline of RCI
Cytopathological classification | Baseline through Week 16 and Week 32
  Change from baseline of cytopathological classification based on bethesda system
Expression rate of P16/Ki-67 | Baseline through Week 16
  Change from baseline as compared to placebo of the expression rate of P16/Ki-67
The number of CD8 positive cells in the cervix | Baseline through Week 16
  Change from baseline as compared to placebo in the number of CD8 positive cells in the cervix
HPV 16 clearance rate | Baseline through Week 16
  Change from baseline as compared to placebo in HPV 16 clearance rate
Change of RCI | Week 16 and Week 32
  Change of RCI based on the histopathological regression at Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Kwan Lee, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (14):
- South Korea (14):
  - Korea University Ansan Hospital, Ansan, Geyonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si, Gyeonggi-do
  - The Dongsan Medical Center of Keimyung Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Yonsei Unversity Health System, Seoul
  - University of Ulsan College of Medicine, Asan Medical Center, Seoul
  - Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Hallym University Medical Center, Seoul
  - Kwandong University College of Medicine Cheil Hospital, Seoul
  - CHA Gangnam Hospital, Seoul
  - Korea University Guro Hospital, Seoul